CLINICAL TRIAL: NCT02610647
Title: Functional Significance of Complexity Measures in the Sensory-motor Behavior: Are There Potential Clinical Applications?
Brief Title: Functional Significance of Complexity Measures in the Sensory-motor Behavior
Acronym: NEURO COMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: LOCAL/2014/ADKT-001; 2014-A01257-40 (Other: ANSM)
Record Dates: First submitted 2015-11-18; First posted 2015-11-20 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2018-01

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control group (Other): Subjects randomized to this group will have a tapping test with no sensory blocking.
  Intervention: Tapping test
  Interventions: Other: Tapping test
- Wrist anesthesia (Experimental): Subjects randomized to this group will have an axillary block / regional anesthesia followed by a tapping test.
  Intervention: Wrist anesthesia
  Intervention: Tapping test
  Interventions: Drug: Wrist anesthesia; Other: Tapping test
- Wrist anesthesia, masked (Experimental): Subjects randomized to this group will have an axillary block / regional anesthesia, will wear a blinding mask, and then will perform a tapping test.
  Intervention: Wrist anesthesia
  Intervention: Blinding mask
  Intervention: Tapping test
  Interventions: Drug: Wrist anesthesia; Other: Blinding mask; Other: Tapping test
- Wrist anesthesia, helmet (Experimental): Subjects randomized to this group will have an axillary block / regional anesthesia, will wear an anti-noise helmet, and then will perform a tapping test.
  Intervention: Wrist anesthesia
  Intervention: Anti-noise helmet
  Intervention: Tapping test
  Interventions: Drug: Wrist anesthesia; Other: Anti-noise helmet; Other: Tapping test
- Wrist anesthesia, masked & helmet (Experimental): Subjects randomized to this group will have an axillary block / regional anesthesia, will wear a blinding mask, will wear an anti-noise helmet, and then will perform a tapping test.
  Intervention: Wrist anesthesia
  Intervention: Blinding mask
  Intervention: Anti-noise helmet
  Intervention: Tapping test
  Interventions: Drug: Wrist anesthesia; Other: Blinding mask; Other: Anti-noise helmet; Other: Tapping test

INTERVENTIONS:
Drug: Wrist anesthesia — Prior to the tapping test, regional anesthesia is performed in the form of sensory blocks distal to the wrist: injection of ropivacaine 7.5mg / ml is carried out successively in contact with three nerves (ulnar, median and radial) with a volume of 2 ml for nerve, for a total of 45mg.
  Arms: Wrist anesthesia; Wrist anesthesia, helmet; Wrist anesthesia, masked; Wrist anesthesia, masked & helmet
Other: Blinding mask — Patients will don a mask that prevents them from seeing during the tapping test.
  Arms: Wrist anesthesia, masked; Wrist anesthesia, masked & helmet
Other: Anti-noise helmet — Patients will don a helmet that prevents them from hearing during the tapping test.
  Arms: Wrist anesthesia, helmet; Wrist anesthesia, masked & helmet
Other: Tapping test — Subjects will be placed at a table in a sitting position where they will perform a rhythmic finger tapping test. The seat height is adjusted so that the front dominant arm rests comfortably on the table. Subjects will be equipped with headphones to receive auditory signals during a first synchronized phase of tapping.
  After the last auditory signal, participants will continue the tapping task by themselves as directed: "after the metronome stops,continue tapping the prescribed tempo as accurately and consistently as possible throughout the test." The movements of the index finger will be measured by a single-axis accelerometer (15 × 15 mm) attached to the nail.

SUMMARY:
The main objective of this study is to compare between groups the level of complexity of the estimated sensorimotor performance through multi-fractal (minmaxMF-DFA) exponents.

DETAILED DESCRIPTION:
The secondary objectives of this study are to compare the level of complexity of the estimated sensorimotor performance using the(A) mono-fractal exhibitors (the αDFA values) and the (B) coefficient of variation (CV) between groups.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The subject does not practice music intensively (<1h / day on average)

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, or under guardianship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient, or breastfeeding
* The subject regularly practices music
* The subject is suffering from a neurodegenerative disease of the central or peripheral nervous system which may affect the sensorimotor control of rhythmic movements of the upper limb
* The subject has had a recent trauma of the upper limb
* The subject is suffering from uncorrected visual and hearing impairment

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
minmaxMF-DFA value during the tapping test | Day 0
  The level of complexity of the estimated sensorimotor performance as measured by the multi-fractal exponents.

SECONDARY OUTCOMES:
Coefficient of variation | Day 0
αDFA value during the tapping test | Day 0
  The level of complexity of the estimated sensorimotor performance as measured by the single-fractal exponent.

CONTACTS AND LOCATIONS:
Overall Officials: Kjerstin Torre, MD, PhD, Study Director — Centre Hospitalier Universitaire de Nîmes
Locations (3):
- France (3):
  - Laboratoire Movement to Health (M2H), Euromov, Université Montpellier 1, Montpellier
  - CHU de Montpellier - Hôpital Lapeyronie, Montpellier
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes

REFERENCES:
- [Result] Torre K, Vergotte G, Viel E, Perrey S, Dupeyron A. Fractal properties in sensorimotor variability unveil internal adaptations of the organism before symptomatic functional decline. Sci Rep. 2019 Oct 31;9(1):15736. doi: 10.1038/s41598-019-52091-y. PMID 31673034